CLINICAL TRIAL: NCT04973566
Title: A Phase 1, Open-Label Study to Investigate Drug-Drug Interaction (DDI) Potential of Nipocalimab With Coadministration of Etanercept or Hydroxychloroquine in Healthy Participants
Brief Title: A Study of Nipocalimab With Co-administration of Etanercept or Hydroxychloroquine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR109053; 2021-001656-33 (EudraCT Number); 80202135EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Etanercept; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Part 1 is a single-sequence, 2-period study and Part 2 is a randomized, 2-cohort (Cohort 1 and Cohort 2), parallel study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Etanercept and Nipocalimab (Experimental): Participants will receive a single subcutaneous (SC) dose of etanercept on Day 1 in Period 1 followed by single intravenous (IV) infusion of nipocalimab on Day 29, SC administration of etanercept followed by an IV infusion of nipocalimab on Day 43 and then a single dose of nipocalimab IV infusion on Day 57 in Period 2 of Part 1. There will be a wash-out period of 28 days between Day 1 of Period 1 and Day 29 of Period 2 in Part 1.
  Interventions: Drug: Nipocalimab; Drug: Etanercept
- Part 2 (Cohort 1): Nipocalimab (Experimental): Participants will receive a single IV infusion of nipocalimab on Day 1 in Cohort 1 of Part 2.
  Interventions: Drug: Nipocalimab
- Part 2 (Cohort 2): Nipocalimab and Hydroxychloroquine (HCQ) (Experimental): Participants will receive a single oral dose of HCQ film-coated tablets once daily from Day 1 to Day 22 and a single IV infusion of nipocalimab on Day 8 in Cohort 2 of Part 2.
  Interventions: Drug: Nipocalimab; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an IV infusion.
  Other Names: JNJ-80202135, M281
Drug: Etanercept — Etanercept will be administered subcutaneously.
  Arms: Part 1: Etanercept and Nipocalimab
Drug: Hydroxychloroquine — HCQ will be administered orally.
  Arms: Part 2 (Cohort 2): Nipocalimab and Hydroxychloroquine (HCQ)

SUMMARY:
The primary purpose of this study is to assess the effect of nipocalimab on the pharmacokinetic (PK) of etanercept (Part 1); and to assess the effect of hydroxychloroquine (HCQ) on total serum immunoglobin G (IgG) reduction by nipocalimab (Part 2) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are any abnormalities, they must be consistent with the underlying illness in the study population or considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening (including immunoglobulin [Ig]G) and at admission to the study site. If the results of the serum chemistry panel, liver panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Good venous access in both arms
* Participants must have heart rate of at least 50 beats per minute
* Participant is considered eligible according to the following tuberculosis (TB) screening criteria (for Part 1 only): a) have no history of latent or active TB before screening; b) have no signs or symptoms suggestive of active TB upon medical history and/or physical examination; c) have had no recent close contact with a person with active TB; d) have a negative QuantiFERON-TB test result within 28 days prior to the administration of study intervention
* Part 1: Body mass index (BMI) greater than or equal to (>=) 18.0 to less than or equal to (<=) 30.0 kilogram (kg)/meter (m)^2 (inclusive), and body weight >= 50 to <= 110.0 kg (inclusive) at the screening visit and on Day -1; Part 2: BMI >= 18.0 to <= 30.0 kg/m^2 (inclusive), and body weight >= 61.5 to <= 110.0 kg (inclusive) at the screening visit and on Day -1
* A female participant must have a negative serum (beta-human chorionic gonadotropin) test at screening and a urine pregnancy test at Day -1 prior to administration of study intervention
* It is recommended that participants are up to date on age-appropriate vaccinations prior to screening per routine local medical guidelines. For study participants who received locally-approved (and including emergency use-authorized) coronavirus disease 2019 (COVID-19) vaccines recently prior to study entry, applicable local vaccine labeling, guidelines, and standards of care for participants receiving immune-targeted therapy should be followed when determining an appropriate interval between vaccination and study enrollment

Exclusion Criteria:

* Has a history of liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has a history of retinal and macular disease (only for Part 2)
* Has shown a previous severe immediate hypersensitivity reaction response, including anaphylaxis, to therapeutic proteins (example, monoclonal antibody [mAbs])
* Has serum albumin levels < 30 grams/Liter (g/L) at screening and Day -1
* Has a history of myocardial infarction, unstable ischemic heart disease, or stroke within 12 weeks prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Part 1: Serum Etanercept Concentration | Up to Day 99
  Serum etanercept concentration will be reported.
Part 1: Ratio of Area Under the Concentration-time Curve (AUCR) of Etanercept | Up to Day 99
  AUCR is defined as the ratio of area under the concentration-time curve.
Part 1: Area Under the Concentration-time Curve of Etanercept from Time Zero to Time of Last Observed Quantifiable Concentration (AUC [0-Last]) | Up to Day 99
  AUC (0-last) is defined as area under the concentration-time curve of etanercept from time zero to time of last observed quantifiable concentration.
Part 1: Area Under the Concentration-time Curve of Etanercept from Time Zero to Infinite time (AUC [0-Infinity]) | Up to Day 99
  AUC (0-Infinity) is defined as area under the concentration-time curve of etanercept from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z) where AUC (0-last) is area under the concentration-time curve of etanercept from time zero to time of last observed quantifiable concentration and C(last) is the last observed quantifiable concentration, and lambda(z) is apparent terminal elimination rate constant.
Part 1: Maximum Observed Concentration (Cmax) of Etanercept | Up to Day 99
  Cmax is defined as maximum observed concentration of etanercept.
Part 1: Ratio of Maximum Observed Concentration (CmaxR) of Etanercept | Up to Day 99
  CmaxR is defined as ratio of maximum observed concentration of etanercept.
Part 1: Time to Reach the Last Observed Measurable Analyte Concentration (Tlast) of Etanercept | Up to Day 99
  Tlast is defined as time to reach the last observed measurable analyte concentration of etanercept.
Part 1: Time to Reach the Maximum Observed Concentration (Tmax) of Etanercept | Up to Day 99
  Tmax is defined as time to reach the maximum observed concentration of etanercept.
Part 1: Elimination Half-life (t1/2) of Etanercept | Up to Day 99
  t1/2 is defined as elimination half-life associated with the terminal slope lambda(z) of the semilogarithmic drug concentration-time curve, calculated as 0.693/ lambda(z).
Part 1: Total Apparent Clearance (CL/F) of Etanercept | Up to Day 99
  CL/F is total apparent clearance of etanercept following subcutaneous (SC) administration, calculated as dose/AUC (0-infinity).
Part 1: Apparent Volume of Distribution (Vdz/F) of Etanercept | Up to Day 99
  Vdz/F is defined as apparent volume of distribution based on the terminal phase after an SC dose, calculated as dose/lambda(z)*AUC(0-infinity).
Part 2: Change from Baseline in Total Serum Immunoglobulin (Ig) Levels | Baseline up to Day 50
  Change from baseline in total serum Ig levels (serum IgG and IgG subtypes) through Day 50 will be reported.

SECONDARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) | Up to 4 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1: Number of Participants with Abnormalities in Physical Examinations | Up to 4 months
  Number of participants with abnormalities in physical examinations (full and brief) will be reported. Full physical examinations will include a review of the following body systems: general appearance; thorough skin and oral mucosa evaluation; eyes, ears, nose, and throat; cardiovascular; respiratory; abdomen; peripheral pulsation; lymph nodes; neurologic; musculoskeletal; head, neck, and thyroid. A brief physical examination includes review of the following body systems: general appearance, thorough skin (including site of the injection) and oral mucosa, abdomen, respiratory, cardiovascular, any abnormalities noted on previous examinations.
Part 1: Number of Participants with Abnormalities in Vital Sign Measurements | Up to 4 months
  Number of participants with abnormalities in vital sign measurements (body temperature [temporal artery measurement], pulse/heart rate, respiratory rate, blood pressure) will be reported.
Part 1: Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 4 months
  Number of participants with abnormalities in clinical laboratory tests (serum chemistry, liver panel, hematology, and urinalysis) will be reported.
Parts 1 and 2: Serum Nipocalimab Concentrations | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  Serum nipocalimab concentrations will be reported.
Part 1: AUCR of Nipocalimab | Up to Day 99
  AUCR is defined as the ratio of area under the concentration-time curve.
Parts 1 and 2: AUC (0-Last) of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  AUC (0-last) is defined as area under the concentration-time curve of nipocalimab from time zero to time of last observed quantifiable concentration.
Parts 1 and 2: AUC (0-Infinity) of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  AUC (0-Infinity) is defined as area under the concentration-time curve of nipocalimab from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z) where AUC (0-last) is area under the concentration-time curve of nipocalimab from time zero to time of last observed quantifiable concentration and C(last) is the last observed quantifiable concentration, and lambda(z) is apparent terminal elimination rate constant.
Parts 1 and 2: Cmax of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  Cmax is defined as maximum observed concentration of nipocalimab.
Part 1: CmaxR of Nipocalimab | Up to Day 99
  CmaxR is defined as ratio of maximum observed concentration of nipocalimab.
Parts 1 and 2: Tlast of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  Tlast is defined as time to reach the last observed measurable analyte concentration of nipocalimab.
Parts 1 and 2: Tmax of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  Tmax is defined as time to reach the maximum observed concentration of nipocalimab.
Parts 1 and 2: t1/2 of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  t1/2 is defined as elimination half-life associated with the terminal slope lambda(z) of the semilogarithmic drug concentration-time curve, calculated as 0.693/ lambda(z).
Parts 1 and 2: Total Systemic Clearance of Nipocalimab (CL) | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  CL is defined as total systemic clearance of nipocalimab following an intravenous (IV) administration, calculated as dose/AUC (0-infinity).
Parts 1 and 2: Volume of Distribution (Vdz) of Nipocalimab | Up to Day 99 (Part 1); up to Day 50 (Part 2)
  Vdz is defined as volume of distribution, based on the terminal phase after an IV dose, calculated as dose/lambda(z)*AUC (0-infinity).
Part 1: Number of Participants with Antibodies to Nipocalimab | Up to Day 99
  Number of participants with antibodies to nipocalimab will be reported.
Part 2: Serum Lipid and Albumin Levels | Up to Day 50
  Participants serum lipid and albumin levels will be reported.
Part 2: Number of Participants with Receptor Occupancy (RO) Levels of Nipocalimab | Up to Day 50
  Number of Participants with RO levels (example, neonatal Fc receptor [FcRn] RO in circulating monocytes) of nipocalimab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency